CLINICAL TRIAL: NCT01853813
Title: First-line FOLFIRI and Bevacizumab in Patients With Advanced Colorectal Cancer Prospectively Stratified According to Serum LDH
Brief Title: First-line Irinotecan, Lederfolin and 5FU (FOLFIRI) and Bevacizumab in Patients With Advanced Colorectal Cancer
Acronym: CENTRAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other)
Collaborators: Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-005048-46
Record Dates: First submitted 2013-03-21; First posted 2013-05-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Colorectal Cancer Stage II
Keywords: colorectal cancer; advanced disease; LDH
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab and FOLFIRI (Other): Bevacizumab 5 mg/kg d1 q14 in combination with FOLFIRI (Irinotecan, leucovorin, 5FU I.V.bolus and 5FU I.V. c.i.)
  Interventions: Drug: Bevacizumab and FOLFIRI

INTERVENTIONS:
Drug: Bevacizumab and FOLFIRI — The CENTRAL trial is a biologically enriched prospective phase II clinical trial in which patients treated with first-line modified FOLFIRI and bevacizumab will be prospectively stratified according to LDH serum levels.
  After written informed consent patients will be enrolled. Patients will be considered evaluable for study aim if response rate was radiologically evaluated at least once during treatment course.
  Treatment will be administered until progression, patients' withdrawal of consent, unacceptable toxicity
  Other Names: CPT11; Folinic acid; 5FU

SUMMARY:
Bevacizumab in combination with chemotherapy represents a standard of care for first-line treatment in patients with advanced colorectal cancer. Molecular predictive factors for bevacizumab efficacy have not yet been identified therefore selection of patients more likely to benefit from such a treatment approach is not possible. Retrospective analyses suggested that LDH serum levels may influence the clinical activity of anti-angiogenetic drugs. Primary aim of our clinical trial will be to prospectively ascertain whether bevacizumab in combination with chemotherapy has an improved clinical activity in patients with high LDH serum levels compared to patients with normal LDH serum levels

DETAILED DESCRIPTION:
The VEGF-driven tumour pathway has been demonstrated to represent a novel therapeutic target for an innovative class of antineoplastic agents. Among these antiangiogenetic-targeted treatment modalities the anti-VEGF monoclonal antibody bevacizumab has become a new standard of care for first-line treatment of metastatic colorectal cancer. The biological link between hypoxia, LDH levels and the tumour-driven angiogenesis pathway through the abnormal activation of the hypoxia Inducible factor 1 α (HIF1-α) is well established. HIF1-α is a key transcription factor that up-regulates a series of genes involved in glycolytic metabolism, angiogenesis, cell survival and erythropoiesis Accordingly to this biological assumption Azuma et al (Azuma et al 2007) demonstrated that high LDH serum levels were associated with tumour over-expression of VEGFA and VEGFR-1. As a clinical consequence it has been speculated that LDH levels may represent an indirect indicator of activated tumour angiogenesis and ultimately of worse prognosis We previously analysed the role of LDH pre-treatment serum levels in colorectal cancer patients receiving first-line bevacizumab in metastatic colorectal cancer treated with first-line bevacizumab were eligible. A control group including all consecutive patients treated with chemotherapy alone was also considered. Pre-treatment LDH serum levels were collected for all cases

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* No prior treatment for advanced disease (adjuvant therapy allowed)
* age < 75 years < 18 years
* Histologically/cytologically confirmed advanced, colorectal cancer
* At least one lesion measurable with CT or MRI scan
* Performance Status (ECOG) 0-1 at study entry)
* Life expectancy of at least 6 months
* Neutrophils count =/> 1.5 x 109/L, platelets count =/> 100 x 109/L, HGB =/> 10 g/dL
* total bilirubin < 1.5 x UNL • SGOT and SGPT =/< 2.5 x UNL (=/< 5 x UNL in patients with liver metastases)
* Creatinine < 1.5 x UNL

Exclusion Criteria:

* CNS metastases
* Severe cardiovascular disease
* Uncontrolled infections
* Radiotherapy within 4 weeks of study entry
* Any experimental drug administered within 4 weeks of study entry
* Known hypersensitivity to study drug
* Known drugs or alcohol abuse
* Pregnant or lactating women (serum Betahcg test)
* Other tumours, except in situ melanoma or cervix cancer if radically removed
* Incapability to sign informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Response Rate | RR will be evaluated every 12 weeks for 24 months
  Response rate to ascertain whether bevacizumab in combination with chemotherapy could determine an improved response rate in patients with high LDH serum levels compared to patients with normal LDH serum levels

SECONDARY OUTCOMES:
Progression free survival | 18 months: time from the start of the treatment until PD or death
  Progression free survival to ascertain whether bevacizumab in combination with chemotherapy could determine an improved progression survival in patients with high serum LDH levels compared to patients with normal LDH serum levels
evaluation of serum IL-8, bFGF, HGF, PlGF, SDF-1, MCP-3 | every 12 weeks for 18 months
  Methods described by Kopetz et al (Kopetz, JCO 2010)

OTHER OUTCOMES:
RECIST criteria and those defined by Chun | every12 weeks for 18 months
  Radiological Criteria defined by Chun (Chun et al, JAMA 2009)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Cascinu, PhD, Study Chair — GISCAD Foundation
Locations (13):
- Italy (13):
  - A.O. Universitaria - Ospedali Riuniti, Ancona, Ancona
  - A.O. Ospedale G.Rummo, Benevento, Benevento
  - A.O. Treviglio-Caravaggio, P.le Ospedale n1, Treviglio, Bergamo
  - Istituto Ospedaliero Fondazione Poliambulanza, Brescia, Brescia
  - Ospedale Civile, Carrara, Massa Carrara
  - Ospedale Maggiore Policlinico, Milan, Milano
  - IRCCS Istituto Europeo di Oncologia, Milan, Milano
  - A.O. Ospedale S.Paolo, Milan, MI
  - Istituto Oncologico Veneto, Padua, PD
  - Ospedale Santa Croce, Fano, PS
  - Azienda Ospedaliera San Carlo, Potenza, PZ
  - Università Policlinico Umberto I, Roma, RM
  - A.O. S.Giovanni Calabita Fatebenefratelli, Roma, Roma